CLINICAL TRIAL: NCT05499403
Title: Treatment fAIlure in Osteoporosis: Who Will Experience a New fRacture? The TAILOR Study
Brief Title: Incidence of the Treatment faIlure in Osteoporosis
Acronym: TAILOR
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Patrizia D'Amelio, associated professor, Centre Hospitalier Universitaire Vaudois
Other Study IDs: TAILOR
Record Dates: First submitted 2022-08-11; First posted 2022-08-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Osteoporosis; Treatment Failure
Keywords: osteoporosis; treatment; fractures
MeSH Terms: conditions — Osteoporosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Osteoporotic fractures are associated with significant morbidity, increased mortality and reduction in the quality of life, available treatments reduces the fracture risk between 30 and 70%, however some patients experience a new fracture and/or continue to loose bone during treatment; this has been defined as treatment failure (TF). The epidemiology and biological bases of TF are currently under-investigated, thus it is impossible for the physician to forecast patients' answer to treatment. The aims of TAILOR study are to collect sounded epidemiological data on TF in a real life setting. To this extent, the investigators will retrospectively a large cohort of 5000 patients with at least 60 months of anti-osteoporotic treatment followed in our center for the diagnosis and care of bone metabolic diseases, and compare TF patients to adequate responders (ARs) for clinical characteristic and biological parameters. The results will be a "signature" to identify those patients who will experience TF.

DETAILED DESCRIPTION:
Fragility fractures represent a major clinical burden in the increasingly older population. Old suffering with femoral fractures will die within a year (15-25%) or become dependent (50%). Costs associated with fractures have been estimated to be 32 billion EUR/year in Europe, 20 billion USD in the United States and 12.5 billion USD in China. The second fracture worsen the patients' health and increases costs, the financial burden imposed by second fractures on the United States healthcare system has been calculated in 2 billion USD/year.

The efficacy of treatment in osteoporosis relies in the reduction of the fracture risk: drugs approved for osteoporosis reduce the risk of fractures between 30-70% for vertebral fractures, 40-50% for hip fractures and 15-20% for non-vertebral fractures (1,2). However, no available treatment reset the fracture risk to zero. Treatment efficacy is assumed by a significant reduction in fracture risk supported by an increase in bone mineral density (BMD) and a decrease in markers of bone turnover. The question if a new fracture or bone loss may be considered a treatment failure is highly debated, recently, a position paper of the International Osteoporosis Foundation described the treatment failure (TF) based on the occurrence of two fractures or one fracture plus lack of variation in BMD, markers of bone turnover or both while on treatment (3).

The study of TF and its prevention is crucial, as the correct and precocious identification of the patients that will not benefit from the first line drugs, will prevent unsuccessful treatment and reduce sanitary costs. Several factors has been suggested to be associated with TF, however, until now, the therapeutic decision relies entirely on physician expertise and not on decisional algorithms.

The aim of this project is to characterize the clinical characteristics foreseeing TF. The identification of a signature for TF will increase the standard care of osteoporotic patients reducing the burden due to a new fracture.

TAILOR will pave the way for the generation of a new algorithm to choose wisely a personalize therapeutical approach for osteoporotic patients, taking into account their clinical characteristics, thus minimizing the risk of TF, improving patients quality and expectancy of life and reducing sanitary costs.

2. Experimental Design and Approach. Retrospective study on patients on treatment with anti-resorptives or anabolics for primary osteoporosis. All the patients evaluated in the out-patients service of the unit between 2009 and 2019 (about 5000 subjects) will evaluated, medical records of patients are available, medical records with missing information will be excluded.

The investigators will include in the analyses women affected by post-menopausal osteoporosis treated for at least 12 months and up to 10 years with drugs active on bone turnover and with at least one follow-up visit in the 10-year period considered. TF will be diagnosed according to the position paper of the IOF (3): occurrence of two fragility fractures while on treatment or one fracture plus lack of variation BMD, biochemical markers or both.

Fragility fracture will be defined because of a fall from the standing position or a mechanical effort without fall. Spinal fractures have be certified by radiography or DXA morphometry whereas for non-vertebral fractures, a hospital discharge or physician report will be also considered valid evidence of fracture. Fractures of the skull, face, cervical spine, fingers, and toes will not be included in our study.

Patients will be considered ARs when they completed 60 months on treatment with no incident fractures according with Diez-Perez et al. (4), for teriparatide the period considered will be 24 months.

Patients will be classified according to the type of drug used (SERMs, oral bisphosphonates, iv bisfosfonates, denosumab or teriparatide), for each patients the following information will be recorded: age, post-menopausal period, assumption of calcium and vitamin D, presence and site of fragility fractures, BMD, serum levels of calcium, phosphate, PTH, creatinine, 25OHvitaminD, markers of bone turnover, adverse events. This information will be recorded at the baseline and at each follow-up visit. The decision of the physician expert in osteoporosis management during the follow-up visit will be recorded (i.d. continue the ongoing treatment or change drug, new drugs prescribed).

Patients will be classified as TF based on the occurrence of two fractures while on treatment or one fracture plus lack of variation in bone mineral density (BMD), biochemical markers or both(3).

Statistical analyses. The power analysis was conducted using an estimated medium effect size (f = 0.25), an alpha level of 0.05, and a power of 0.95 using the software G*power. According to statistical computing, a sample size of n = 400 is required.

The percentage of TF within different treatment and will be compared with AR by means of ANCOVA for analyzed variables.

the medical decision taken by the physician expert in bone metabolic disorders after treatment failure (the patient will continue the treatment/switch to another treatment/stop treatment) will be analysed.

References

1. Body J-J, Bergmann P, Boonen S, Boutsen Y, Devogelaer J-P, Goemaere S, Kaufman J-M, Rozenberg S, Reginster J-Y. Evidence-based guidelines for the pharmacological treatment of postmenopausal osteoporosis: a consensus document by the Belgian Bone Club. Osteoporos Int. 2010 Oct;21(10):1657-80.
2. MacLean C, Newberry S, Maglione M, McMahon M, Ranganath V, Suttorp M, Mojica W, Timmer M, Alexander A, McNamara M, Desai SB, Zhou A, Chen S, Carter J, Tringale C, Valentine D, Johnsen B, Grossman J. Systematic review: comparative effectiveness of treatments to prevent fractures in men and women with low bone density or osteoporosis. Ann Intern Med. 2008 Feb 5;148(3):197-213.
3. Diez-Perez A, Adachi JD, Agnusdei D, Bilezikian JP, Compston JE, Cummings SR, Eastell R, Eriksen EF, Gonzalez-Macias J, Liberman UA, Wahl DA, Seeman E, Kanis JA, Cooper C, IOF CSA Inadequate Responders Working Group. Treatment failure in osteoporosis. Osteoporos Int. 2012 Dec;23(12):2769-74.
4. Díez-Pérez A, González-Macías J. Inadequate responders to osteoporosis treatment: proposal for an operational definition. Osteoporos Int. 2008 Nov;19(11):1511-6.

ELIGIBILITY:
Inclusion Criteria:

* patients affected by post-menopausal osteoporosis
* patients treated for at least 12 months and up to 10 years with drugs active on bone turnover
* patients with at least one follow-up visit in the period considered by the study

Exclusion Criteria:

* male gender
* glucocorticoid use (more than 3 months at any time)
* metabolic or endocrine disease with bone effect
* prolonged immobilization (patients not able to walk independently for more than 3 months at any time)
* chronic gastrointestinal disease (eg, resection or derivative surgery, inflammatory bowel disease)
* malabsorption
* multiple myeloma
* chronic obstructive pulmonary disease
* renal failure (estimated glomerular filtration rate [GFR]<30 mL/min).

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Patients on treatment with anti-resorptives or anabolics for primary osteoporosis. We will include in the analyses all the patients evaluated in the out-patients service of our unit between 2009 and 2019 (about 5000 subjects), medical records of patients are available, medical records with missing information will be excluded.
  TF will be diagnosed according to the position paper of the IOF: occurrence of two fragility fractures while on treatment or one fracture plus lack of variation BMD, biochemical markers or both.
Sampling Method: Non-Probability Sample
Enrollment: 415 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
incidence of treatment failure (TF) | 60 months
  incidence of TF for different type of drugs used in osteoporosis.

SECONDARY OUTCOMES:
risk factors (odds ratio) | 60 months
  risk factors for treatment failure

CONTACTS AND LOCATIONS:
Locations (1):
- Patrizia D'amelio, Lausanne, Switzerland